CLINICAL TRIAL: NCT03199417
Title: Trial Evaluating multimOdal toPical Cream In CompArison to pLacebo (TOPICAL)
Acronym: TOPICAL
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Terminated prematurely due to feasibility issues with rate of recruitment
Sponsor: University of Michigan (Other)
Collaborators: McMaster University (Other); Oakville Trafalgar Memorial Hospital (Unknown)
Responsible Party: Principal Investigator, Neil Bakshi, Researcher, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017/02
Record Dates: First submitted 2017-06-21; First posted 2017-06-26 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Single center blinded randomized controlled trial with a random number generator determining the allocation of patients to either the placebo or intervention groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized using a random number generator to either intervention. Interventions will be identically packaged and labeled either A or B by a pharmacist who will be uninvolved with the trial administration. Participants and study personnel will be blinded to the treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiprofen/interventional (Experimental): A multimodal topical cream treatment with Ketoprofen, Baclofen, Amitryptiline, and lidocaine in a carrier gel. This topical formulation has been in use commercially under the trade name "Multi-profen". This topical cream will be applied by the patient three times per day.
  Interventions: Drug: Multiprofen
- Control/Placebo Group (Placebo Comparator): A identically packaged placebo cream treatment will be utilized in the control population.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Multiprofen — A multimodal topical cream treatment with Ketoprofen, Baclofen, Amitryptiline, and lidocaine in a carrier gel.
  Arms: Multiprofen/interventional
Other: Placebo — An identically packaged placebo cream
  Arms: Control/Placebo Group

SUMMARY:
Randomized controlled trial regarding the efficacy of a multimodal topical analgesic, Multiprofen, in comparison to placebo cream treatment on knee pain and function in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a disease with a high global burden, and multiple conservative treatment options are available. In addition to being a major source of disability osteoarthritis results in a significant economic burden as well. A study published in 2012 showed the 1-year physician, outpatient procedure, and hospitalization costs in patients with osteoarthritis more than double those patients without osteoarthritis in Ontario.

Conservative treatment options include topical and oral anti-inflammatory medications, weight loss, physiotherapy and intra articular cortisone and viscosupplementation injections. Unfortunately, commonly used treatments such as oral anti-inflammatory medications carry a significant systemic adverse effect on the gastrointestinal (GI) tract and hepatic and renal systems and intra articular cortisone have potential adverse effect on blood glucose control. For this reason, topical anti-inflammatory medications are popular yet are often ineffective. Unfortunately, topical anti-inflammatory medications have variable efficacy in relieving osteoarthritic knee pain and often only provide a moderate degree of pain relief.

In the setting of chronic pain various other topical modalities have been utilized. A systematic review of the literature identified commonly studied topical analgesics were nonsteroidal anti-inflammatory drugs followed by lidocaine, capsaicin, amitriptyline, glyceryl trinitrate, opioids, menthol, pimecrolimus, and phenytoin. Given the biological bases behind utilizing agents which target a variety of pain generators the investigators hypothesized that a combination of these would provide significant pain relief to patients affected by end stage knee osteoarthritis. For this reason, the investigators propose a trial evaluating utilizing multiple topical modalities for pain relief to provide support for the use of combination therapy in treating knee osteoarthritis. Results from this study will potentially improve the global health and economic burden through improvement in the management of knee osteoarthritis.

STUDY OBJECTIVES

Primary objective The primary objective of the trial will be to evaluate the efficacy of a multimodal topical analgesic, Multiprofen, in comparison to placebo cream treatment on patient reported pain relief utilizing a 11-point visual analog scale (VAS) measured from 0-10.

Secondary objectives

Our secondary objectives will be to evaluate the effect of topical combination therapy on:

1. Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) patient reported outcome score. This score is commonly utilized in assessment of knee osteoarthritis and has been validated to be reliable and responsive in this patient population.
2. Patient knee range of motion and strength
3. Return to previous level of activity
4. Radiographic degree of osteoarthritis.
5. Patient demographics
6. Adverse events

SUMMARY OF TRIAL DESIGN The investigators propose a single center blinded trial evaluating the efficacy of a combination formula of topical analgesic in comparison to placebo cream treatment. The investigators will randomize 186 patients between topical multimodal cream "multiprofen" and a control placebo cream.

Randomization Method Participants will be randomized using a random number generator to either experimental or placebo control intervention.

Participants will be randomized to one of two treatments:

Experimental - A multimodal topical cream treatment with Ketoprofen, Baclofen, Amitryptiline, and lidocaine in a carrier gel. This topical formulation has been in use commercially under the trade name "Multi-profen".

Control - A identically packaged placebo cream treatment will be utilized in the control population.

Proposed duration of treatment and follow-up: Participants will be brought back at 3,6 and 12 weeks' time to complete questionnaires recording VAS and WOMAC scores

The current proposal includes 1 clinical site in Canada (Oakville Trafalgar Memorial Hospital, Oakville, ON, CAN)

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria are:

1. adult men or women ages 50-80 years;
2. Diagnosis of symptomatic osteoarthritis of the knee based on clinical and radiographic criteria;
3. provision of informed consent.

Exclusion Criteria:

The exclusion criteria are:

1. patients with inflammatory osteoarthritis;
2. open wounds or sores over the knee joint;
3. patients that will likely have problems, in the judgment of the investigators, with maintaining follow-up;
4. Cases involving litigation.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Change in pain visual analog scale (VAS) scores (0-10) from baseline | week 0, week 3, week 6, week 12
  Measurement of change in patient reported pain score (VAS) at various follow up appointments. The scale is from 0-10, with 10 being the most pain.

SECONDARY OUTCOMES:
Change in Western Ontario and McMaster Universities Arthritis Index (WOMAC) scores from baseline | week 0, week 3, week 6, week 12
  Change in patient reported knee pain and function scores. WOMAC score has 3 subdivisions which include knee pain, stiffness, and physical function. The score ranges from 0-96, with lower scores representing better knee pain, stiffness, and function.
Change in Range of motion (ROM) from baseline | week 0, week 3, week 6, week 12
  Change in range of motion of the knee at various time points that will be compared to pre-treatment range of motion. Higher range of motion is correlated with better outcome and better function.

CONTACTS AND LOCATIONS:
Overall Officials: Moin Khan, MD, Principal Investigator — MCMASTER
Locations (1):
- Oakville Trafalgar Memorial Hospital, Oakville, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tarride JE, Haq M, O'Reilly DJ, Bowen JM, Xie F, Dolovich L, Goeree R. The excess burden of osteoarthritis in the province of Ontario, Canada. Arthritis Rheum. 2012 Apr;64(4):1153-61. doi: 10.1002/art.33467. Epub 2011 Nov 11. PMID 22081470
- [Background] Rannou F, Pelletier JP, Martel-Pelletier J. Efficacy and safety of topical NSAIDs in the management of osteoarthritis: Evidence from real-life setting trials and surveys. Semin Arthritis Rheum. 2016 Feb;45(4 Suppl):S18-21. doi: 10.1016/j.semarthrit.2015.11.007. Epub 2015 Dec 2. PMID 26806189
- [Background] Stanos SP, Galluzzi KE. Topical therapies in the management of chronic pain. Postgrad Med. 2013 Jul;125(4 Suppl 1):25-33. doi: 10.1080/00325481.2013.1110567111. PMID 24547601
- [Background] Argoff CE. Topical analgesics in the management of acute and chronic pain. Mayo Clin Proc. 2013 Feb;88(2):195-205. doi: 10.1016/j.mayocp.2012.11.015. PMID 23374622
- [Background] Williams VJ, Piva SR, Irrgang JJ, Crossley C, Fitzgerald GK. Comparison of reliability and responsiveness of patient-reported clinical outcome measures in knee osteoarthritis rehabilitation. J Orthop Sports Phys Ther. 2012 Aug;42(8):716-23. doi: 10.2519/jospt.2012.4038. Epub 2012 Mar 8. PMID 22402677
- [Background] Katz NP, Paillard FC, Ekman E. Determining the clinical importance of treatment benefits for interventions for painful orthopedic conditions. J Orthop Surg Res. 2015 Feb 3;10:24. doi: 10.1186/s13018-014-0144-x. PMID 25645576
- [Background] Jabbari M, Hashempur MH, Razavi SZ, Shahraki HR, Kamalinejad M, Emtiazy M. Efficacy and short-term safety of topical Dwarf Elder (Sambucus ebulus L.) versus diclofenac for knee osteoarthritis: A randomized, double-blind, active-controlled trial. J Ethnopharmacol. 2016 Jul 21;188:80-6. doi: 10.1016/j.jep.2016.04.035. Epub 2016 Apr 26. PMID 27125590
- [Result] Fernandez-Lopez JC, Laffon A, Blanco FJ, Carmona L; EPISER Study Group. Prevalence, risk factors, and impact of knee pain suggesting osteoarthritis in Spain. Clin Exp Rheumatol. 2008 Mar-Apr;26(2):324-32. PMID 18565256